CLINICAL TRIAL: NCT04002180
Title: Specified Drug-Use Survey on Entyvio for IV Infusion 300 mg [Crohn's Disease]
Brief Title: Specified Drug-Use Survey on Vedolizumab for IV Infusion 300 mg [Crohn's Disease]
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4021; jRCT1080224753 (Registry Identifier: jRCT)
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Infusions, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vedolizumab 300 mg: Vedolizumab (Genetical Recombination) 300 mg, IV infusion, at Weeks 0, 2 and 6, and every 8 weeks thereafter, for up to 54 weeks. Participants will receive IV infusion as part of routine medical care.
  Interventions: Drug: Vedolizumab (Genetical Recombination)

INTERVENTIONS:
Drug: Vedolizumab (Genetical Recombination) — Vedolizumab IV infusion
  Other Names: Entyvio for IV Infusion 300 mg

SUMMARY:
The purpose of this survey is to evaluate the long-term safety and effectiveness of vedolizumab for intravenous (IV) infusion 300 milligrams (mg) in Crohn's disease (CD) patients in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called vedolizumab for IV infusion 300 mg. This drug is being tested to treat patients who have CD.

This survey is an observational (non-interventional) study and will look at the long-term safety and effectiveness of vedolizumab for IV infusion 300 mg in the routine clinical setting. The planned number of observed patients will be approximately 300.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Have moderate or severe active CD
2. Have inadequate response to existing therapies

Exclusion Criteria:

Patients with any contraindication for vedolizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CD patients treated with vedolizumab for IV infusion 300 mg as part of routine medical care
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who have One or More Adverse Events | Up to Week 54
  Adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Number of Participants who have One or More Adverse Drug Reactions | Up to Week 54
  AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.

SECONDARY OUTCOMES:
Change from Baseline in Crohn's Disease Activity Index (CDAI) Score | Baseline and after 3 doses of vedolizumab (Week 6 to 14), and Week 54 (or discontinuation of vedolizumab therapy)
  CDAI is scoring system for the assessment of Crohn's Disease Activity. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Percentage of Participants with CDAI-100 Response | Baseline and after 3 doses of vedolizumab (Week 6 to 14), and Week 54 (or discontinuation of vedolizumab therapy)
  CDAI-100 response is defined as ≥100-point decrease from baseline in the CDAI score. CDAI is scoring system for the assessment of Crohn's Disease Activity. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Percentage of Participants with CDAI-70 Response | Baseline and after 3 doses of vedolizumab (Week 6 to 14), and Week 54 (or discontinuation of vedolizumab therapy)
  CDAI-70 response is defined as ≥70-point decrease from baseline in the CDAI score. CDAI is scoring system for the assessment of Crohn's Disease Activity. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Percentage of Participants with Clinical Remission | Baseline and after 3 doses of vedolizumab (Week 6 to 14), and Week 54 (or discontinuation of vedolizumab therapy)
  Clinical remission is defined as CDAI score of ≤150 points. CDAI is scoring system for the assessment of Crohn's Disease Activity. Index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Change from Baseline in Quality of Life (QOL) Assessment using Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Baseline and after 3 doses of vedolizumab (Week 6 to 14), and Week 54 (or discontinuation of vedolizumab therapy)
  The SIBDQ is an instrument used to assess quality of life and is a disease-specific health-related quality of life questionnaire, that consists of 10 questions, each question is scored on a scale from 1 (poor quality of life) to 7 (good quality of life). The total score will be reported and is ranging from 10 to 70 with a higher score indicates a better health-related quality of life.
Change from Baseline in White Blood Cell Count | Baseline and up to Week 54
Change from Baseline in Lymphocytes | Baseline and up to Week 54
Change from Baseline in Hemoglobin | Baseline and up to Week 54
Change from Baseline in Hematocrit | Baseline and up to Week 54
Change from Baseline in Albumin | Baseline and up to Week 54
Change from Baseline in C-reactive protein (CRP) | Baseline and up to Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a339